CLINICAL TRIAL: NCT07037966
Title: Truly Portable MRI for Extremity and Brain Imaging Anywhere & Everywhere
Brief Title: Advancing Portable Brain Imaging: The NextMRI Project's Role in Revolutionizing Diagnostic MRI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Collaborators: National Research Council, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NextMRI Brain Validation
Record Dates: First submitted 2025-05-20; First posted 2025-06-26 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; MRI; Brain Imaging
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: All participants receive the same intervention. There's no randomization.-the aim is to evaluate the performance of the device within the same group of patients.
Masking Description: The radiologist is assessing the diagnostic outcome without knowledge of the reference scan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Suspected Multiple Sclerosis (Experimental): A total of 50 patients aged between 18 and 65 years with suspected multiple sclerosis will be scanned using both the 3T MRI and the NextMRI prototype.
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — Standard 3T MRI Scan
Device: MRI — Low-field MRI scan using the NextMRI prototype

SUMMARY:
Mobile imaging diagnostic devices are extremely valuable for clinical diagnosis both inside and outside healthcare facilities. However, Magnetic Resonance Imaging (MRI)-the gold standard for diagnosing many neurological and musculoskeletal conditions-is not easily portable. Moreover, due to its high cost (in the million-euro range) and limited availability, the average wait time in Europe for an MRI scan is from several weeks to months.

The NextMRI project aims to take the technical, industrial, and commercial steps required to deploy portable low-field MRI systems in remote and developing regions, rural areas, sporting events, military or medical camps, and home healthcare settings, improving diagnostic capabilities. The specific goals of the NextMRI project are:

1. Expand current low-field MRI technology to brain imaging.
2. Enhance diagnostic accuracy using machine learning.
3. Improve portability and usability for end users.
4. Reduce production costs for broader affordability.
5. Collect clinical evidence through trials to validate medical performance.
6. Develop a sustainable business model for market commercialization.

DETAILED DESCRIPTION:
Based on this context, the NextMRI project will carry out a clinical evaluation study involving a multidisciplinary team of radiologists, rheumatologists, physiotherapists, data managers, and physicists. The study will focus on patients with suspected multiple sclerosis (MS). Its main goals are to:

1. Assess the diagnostic value of the low-field MRI prototype.
2. Evaluate usability for end users.
3. Train AI algorithms using deep learning to differentiate between healthy and damaged tissues, thereby aiding radiologists, reducing diagnostic time, and lightening their workload.

Radiologists will first generate structured reports based on standard high-resolution MRI scans. They will then evaluate the low-field MRI images from the NextMRI prototype. The initial high-field MRI reports will serve as the reference standard for assessing performance and training the AI system.

Each patient will undergo two MRI scans on the same day (after providing informed consent): one at the standard 3T MR scan and other at the low-field MRI scan (NextMRI). To prevent bias, both scans will be interpreted by a professional radiologist with an 8-week interval between readings.

A total of 50 patients aged between 18 and 65 years with suspected multiple sclerosis will be included. Patients with any contraindications for high-field MRI will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected multiple sclerosis

Exclusion Criteria:

* Any contradictions for high-field MRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Radiological reports to Evaluate NextMRI prototype performance | Through study completion, an average of 1 year
  A clinical evaluation study will be performed involving a multidisciplinary team of radiologists, traumatologists, rheumatologists, physiotherapists, data managers and physicists.
  The validation strategy will be structured in 3 steps:
  1. Radiologists will report the high-resolution MR images in a structured report as part of their clinical duties.
  2. Radiologists will evaluate the MR images acquired with the PR Gen III scanner after 8 weeks, in order be blind to the first reading and avoid learning interobserver bias
  3. Finally, the gold standard information obtained by the initial radiological report will serve to evaluate the prototype performance and train the Deep Learning tools.
  The report documents technical details, contrast use, and lesion analysis in brain, spine, and medulla. It quantifies key MS-related lesions, categorizes locations, and notes other abnormalities. A diagnostic impression summarizes findings to support MS diagnosis.

SECONDARY OUTCOMES:
Patient Comfort and Satisfaction Questionnaire to Evaluate the New NextMRI Prototype Compared to the Standard MRI Scanner | 1 year
  Patients provide insights into their experiences with both scanners, focusing on aspects such as ease of entry and exit, comfort during positioning, perception of claustrophobia, noise levels, and overall satisfaction. Additionally, they compare the two scanners directly, offering valuable perspectives on which device they prefer and why. Their comments highlight subjective comfort and practical challenges, which are critical for improving patient-centered design.
  The Questionnaire will use a Likert scale (e.g., from 1 = very uncomfortable to 5 = very comfortable) combined with open-ended questions for additional comments.
User Comfort and Satisfaction Questionnaire Evaluate the New NextMRI Prototype Compared to the Standard MRI Scanner | 1 year
  Healthcare professionals, including radiologists and MRI technicians, evaluate the scanners from an operational standpoint. Their feedback covers ease of use, image quality, workflow efficiency, technical issues, and overall satisfaction with the device's performance. They also compare the NextMRI prototype to the standard scanner, assessing its potential impact on clinical practice, particularly for patients with conditions like Multiple Sclerosis. Professionals are asked to identify any anticipated challenges in implementation and to suggest additional training or resources needed for optimal use.
  The Questionnaire will use a Likert scale (e.g., from 1 = very uncomfortable to 5 = very comfortable) combined with open-ended questions for additional comments.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario y Politécnico la Fe, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guallart-Naval T, Algarin JM, Pellicer-Guridi R, Galve F, Vives-Gilabert Y, Bosch R, Pallas E, Gonzalez JM, Rigla JP, Martinez P, Lloris FJ, Borreguero J, Marcos-Perucho A, Negnevitsky V, Marti-Bonmati L, Rios A, Benlloch JM, Alonso J. Portable magnetic resonance imaging of patients indoors, outdoors and at home. Sci Rep. 2022 Jul 30;12(1):13147. doi: 10.1038/s41598-022-17472-w. PMID 35907975
- [Background] O'Reilly T, Teeuwisse WM, de Gans D, Koolstra K, Webb AG. In vivo 3D brain and extremity MRI at 50 mT using a permanent magnet Halbach array. Magn Reson Med. 2021 Jan;85(1):495-505. doi: 10.1002/mrm.28396. Epub 2020 Jul 5. PMID 32627235
- See also: Truly portable MRI for extremity and brain imaging anywhere & everywhere — https://nextmri.eu/